CLINICAL TRIAL: NCT03858894
Title: A Randomized, Double-Masked, Parallel-Group, Multicenter Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution 0.002% Once Daily and Twice Daily in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension SPECTRUM 6 Study.
Brief Title: Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution Once Daily and Twice Daily in Subjects With Primary Open-Angle Glaucoma SPECTRUM 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011712IN
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Primary Open-angle Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Arm: DE-117 QD (Experimental): DE-117 Ophthalmic Solution QD (20:00) and Vehicle (8:00; no active DE-117 ingredient) QD
  Interventions: Drug: DE-117 Ophthalmic Solution QD
- Test Arm: DE-117 BID (Experimental): DE-117 Ophthalmic Solution BID Twice daily (20:00 and 8:00)
  Interventions: Drug: DE-117 Ophthalmic Solution BID

INTERVENTIONS:
Drug: DE-117 Ophthalmic Solution QD — DE-117 ophthalmic solution QD and Vehicle (no active DE-117 ingredient) QD add one drop in each eye
  Arms: Drug Arm: DE-117 QD
Drug: DE-117 Ophthalmic Solution BID — DE-117 ophthalmic solution BID twice Daily (20:00 and 8:00) add one drop in each eye
  Arms: Test Arm: DE-117 BID

SUMMARY:
This is a randomized, double-masked, parallel-group, multi-center study. Subjects diagnosed with POAG or OHT who meet eligibility criteria at Visit 1 (Screening) will wash out their current topical IOP lowering medication(s), if any. After completing the required washout period, subjects will return for Visit 2 (Baseline, Day 1). Subjects who meet all eligibility criteria at Visit 2 (Baseline, Day 1) will be randomized to receive study medication for up to 6 weeks.

Approximately 100 subjects with POAG or OHT will be randomized in a 1:1 ratio to either:

* DE-117 ophthalmic solution 0.002% QD (Once Daily)
* DE-117 ophthalmic solution 0.002% BID (Twice Daily)

This study will consist of a screening period of up to 35 days including a washout period of up to 28 days (+ 7 days window), and a 6-week double-masked treatment period.

ELIGIBILITY:
Inclusion Criteria:

Provide signed written informed consent

* Have a diagnosis of POAG or OHT in both eyes, or one eye with POAG and the other with OHT.
* Qualifying corrected visual acuity in each eye
* Qualifying central corneal thickness in each eye
* Qualifying Day 1 IOP measurement at 3 time-points in both eyes
* Qualifying Anterior chamber angle

Exclusion Criteria:

* History of ocular surgery specifically intended to lower IOP
* Subjects who cannot safely discontinue use of ocular hypotensive medications during the wait/washout period
* Advanced glaucoma in either eye
* Any corneal abnormality or other condition interfering with or preventing reliable Goldmann applanation tonometry
* Any ocular surgery or ocular laser treatment within 180 days prior to Screening and throughout the study in either eye
* Females who are pregnant, nursing, or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - East West Eye Institute, Los Angeles, California
  - Danbury Eye Specialist, Danbury, Connecticut
  - Hernando Eye Institute, Brooksville, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Tekwani Vision Center, St Louis, Missouri
  - Eye Associates/SurgiCenter of Vineland, Vineland, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Apex Eye Clinical Research, LLC, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Scott & Christie and Associates PC, Cranberry Township, Pennsylvania
  - University Eye Specialist, Maryville, Tennessee
  - Advanced Vision Research, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Started | 48 | 50
Completed | 44 | 50
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.45) | 66.3 (8.73) | 66.8 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 21 | 25 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 46 | 48 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 14 | 27
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Week 2
Description: Intraocular pressure (IOP), the fluid pressure inside the eye, was measured by applanation tonometry in millimeters mercury (mmHg).
Time Frame: 08:00 at week 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 18.19 (0.46) | 19.15 (0.45)

2. Primary Outcome: Intraocular Pressure (IOP) at Week 2
Description: as for outcome 1
Time Frame: 12:00 at week 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 17.73 (0.49) | 18.17 (0.46)

3. Primary Outcome: Intraocular Pressure (IOP) at Week 2
Description: Intraocular pressure (IOP), the fluid pressure inside the eye, was mea...
Time Frame: 16:00 at week 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 16.73 (0.47) | 17.81 (0.44)

4. Primary Outcome: Intraocular Pressure (IOP) at Week 6
Description: as for outcome 1
Time Frame: 08:00 at week 6
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 18.33 (0.49) | 19.01 (0.47)

5. Primary Outcome: Intraocular Pressure (IOP) at Week 6
Description: as for outcome 1
Time Frame: 12:00 at week 6
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 17.77 (0.45) | 18.35 (0.43)

6. Primary Outcome: Intraocular Pressure (IOP) at Week 6
Description: Intraocular pressure (IOP), the fluid pressure inside the eye, was mea...
Time Frame: 16:00 at week 6
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 17.30 (0.45) | 17.66 (0.43)

7. Secondary Outcome: Mean Diurnal Intraocular Pressure (IOP)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
Number analyzed (Participants) | 48 | 50
mmHg | 17.77 (0.43) | 18.37 (0.41)

ADVERSE EVENTS:
Time Frame: All SAEs were collected from the signing of the Inform Consent Form until the subject withdrew or completed the scheduled exit visit at Week 6.
Arm/Group | Test Arm: DE-117 BID | Drug Arm: DE-117 QD
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/50
Other Adverse Events (participants affected / at risk) | 20/48 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Arm: DE-117 BID (N=48) | Drug Arm: DE-117 QD (N=50)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Arm: DE-117 BID (N=48) | Drug Arm: DE-117 QD (N=50)
Conjunctival hyperaemia (Eye disorders) | 6 (7) | 0 (0)
Ocular hyperaemia (Eye disorders) | 5 (5) | 1 (1)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0)
Corneal pigmentation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Glare (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1)
Vital dye staining cornea present (Investigations) | 2 (3) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site/Investigator is not permitted to publish results communications without Santen's consent until after a period of sixty (60 days) for Santen review/comment. Santen may request removal of any Confidential Information (other than Study results) from manuscripts or materials prior to submission or presentation. At Santen's request Site/Investigator has to withhold any publication if there is a patentable invention until such time as Santen is able to secure adequate patent protection.

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03858894/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03858894/SAP_001.pdf